CLINICAL TRIAL: NCT07047495
Title: MINIONS - Patient-specific Microstructural and radIobiological Model for persoNalised External Beam radiatION Therapy in Localised tumourS
Brief Title: Personalization of External Beam Radiation Therapy in Localised Tumours
Acronym: MINIONS
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: UID 4631
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2024-10

CONDITIONS: Breast Adenocarcinoma; Prostate Cancer (Adenocarcinoma)
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Within the prospective study, biological specimens from patients undergoing in-room biopsy before RT, will be collected. Histological evaluation and cell culture (and organoid preparation) will be conducted, and samples/organoids will be irradiated with RT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prostate patients: prostate patients undergoing RT
  Interventions: Other: prostate patient
- breast patients: breast patients undergoing RT
  Interventions: Other: breast patients

INTERVENTIONS:
Other: prostate patient — patients with prostate cancer treated with RT at IEO
  Groups: Prostate patients
Other: breast patients — patients with breast cancer treated with RT at IEO
  Groups: breast patients

SUMMARY:
The study will include the prospective acquisition of optimized MR imaging data of prostate and breast patients treated with radiotherapy (RT).

Within the prospective study, biological specimens from patients undergoing in-room biopsy before RT, will be collected. Histological evaluation and cell culture (and organoid preparation) will be conducted, and samples/organoids will be irradiated with RT for biological validation.

ELIGIBILITY:
Inclusion criteria for prostate patients:

* Unifocal infiltrating ductal breast carcinoma, non-special histotype
* clinical stage T1-T2,N0
* No contraindications to MRI, or metal joint prostheses from knee to shoulder included, or femoral stent.
* Patients aged >18 years
* Good general condition (ECOG 0-2)
* Expected active treatment (crioablation or surgery or radiotherapy ).

Exclusion Criteria:

* Exclusion criteria for prostate patients:

  * Nodule involvement and metastasis (cN1 and/or cM1)
  * Concomitant inflammation of the intestine
  * Significant systemic diseases or ongoing oral anticoagulant therapy
  * Non-compliance of dose constraints in the treatment plan
  * Previous invasive cancer, unless the patient has had no disease for at least 3 years
  * Mental disorders that cannot ensure valid informed consent

Exclusion criteria for breast patients:

* Histology other than non-special histotype and non-epithelial tumors (sarcoma, lymphoma)
* Male sex
* High-risk mutation carrier patients
* Bilateral breast cancer
* synchronous distant metastases
* Neoadjuvant therapy
* autoimmune connective tissue diseases
* previous radiotherapy to the chest
* Mental disorders that cannot ensure valid informed consent
* No previous thoracic radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include prostate and breast patients undergoing RT.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Generation of in-silico tumor model | 1 year
  generate an in-silico tumour model able to describe tumour microstructure and its interaction with the radiation beam
Personalization of the tumour model with patient-specific MR imaging data | 1 year
  personalize the tumour model implemented in A1 with patient-specific MR imaging data for tumour characterization and treatment outcome prediction, relying on retrospective data
Improvement of personalized tumor-models | 3 years
  Improvement of the implemented models, by relying on advanced agnetic Resonance Imaging (MRI) data acquired prospectively
Evaluation of tumor model in describing the in-vivo microstructural and radiobiological characteristics | 3 years
  The evaluation of the implemented in-silico tumour model in describing the in-vivo microstructural and radiobiological characteristics, by collecting histopathological features and irradiating primary cell cultures.

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Marvaso, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy, Italy